CLINICAL TRIAL: NCT00615862
Title: Relationship Between Alcohol Use Disorders and Cortisol Levels in Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM11399
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2009-06

CONDITIONS: Sepsis; Alcoholism
Keywords: Sepsis, alcoholism, cortisol, delirium, critical care
MeSH Terms: conditions — Sepsis; Alcoholism; Delirium | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Diagnosis of alcohol use disorders will be made through the use of a validated questionnaire.
  2. Blood collected as part of routine patient care (and that is destined to be discarded) will be evaluated for a number of immune markers. Cortisol levels measured as part of routine care will be recorded.
  3. Delirium will be assessed through the use of a validated instrument.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AUD+ and AUD-: AUD stands for alcohol use disorders. Patients with alcohol use disorders are assigned the label AUD+. Patients without alcohol use disorders are assigned the label AUD-.
  Interventions: Other: Observational study; no interventions

INTERVENTIONS:
Other: Observational study; no interventions — Validated questionnaires will be administered. Blood samples will be analyzed for levels of immune markers as well as cortisol. This is an observational study and patients will not undergo any treatment as part of study participation. Patients will not receive medications or other interventions if they participate in the study. Blood samples analyzed are from samples remaining in the hospital laboratory that were collected as part of routine patient care and destined to be discarded.

SUMMARY:
Patients with alcohol use disorders are often cared for in the intensive care unit (ICU). We estimate that close to half of the patients we care for in our ICU have alcohol use disorders. One of the reasons that patients with alcohol use disorders are frequently cared for in our ICU is because patients with alcohol use disorders are at higher risk of developing infections. The medical term for infections is sepsis. When an infection develops, patients with alcohol use disorders tend to get more severely ill compared to patients who do not have alcohol use disorders. Patients with alcohol use disorders are also at higher risk of dying when they develop severe infections.

The purpose of this study is to determine why patients with alcohol use disorders become more severely ill when they develop infections. There are a number of reasons why this is possible. One reason is that a hormone called cortisol is higher in individuals with alcohol use disorders (who do not have infections). This hormone is also higher in patients who are at increased risk of dying from severe infections. One of the aims of this study is to see if cortisol levels are higher in patients with alcohol use disorders compared to those who do not have alcohol use disorders.

Another reason why patients with alcohol use disorders are at increased risk of developing infections is because their immune system is not functioning properly. A second aim of this study is to see if certain markers of immune function are different in patients with alcohol use disorders compared to patients without alcohol use disorders.

Patients with alcohol use disorders are also more likely to become confused when they are in the ICU. This condition is called delirium. Delirium is marked by abrupt onset of altered level of consciousness, disorganized thinking, and inattention that changes over time. Delirium tremens is one form of delirium. About 80% of our ICU patients develop delirium, and many patients who do not have alcohol use disorders develop the disorder as well. Patients with alcohol use disorders who have high cortisol levels have a higher chance of developing delirium compared to patients with normal cortisol levels. A third aim of this study is to examine the relationship between delirium and cortisol in both patients with and without alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the medical intensive care unit at Virginia Commonwealth University Medical Center (also known as Medical College of Virginia Hospitals) in Richmond, Virginia

Exclusion Criteria:

Study exclusion criteria are:

* Age < 18 years old
* Prisoners under legal coercion or restriction
* Pregnant women
* Admission diagnosis other than sepsis
* Admitted to the medical intensive care unit service from location other an emergency department
* No cortisol level measured by the pathology laboratory at Virginia Commonwealth University Medical Center within the first 24 hours after presentation to an emergency department; AND
* Administration of etomidate within 24 hours prior to measurement of cortisol levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the medical intensive care unit at Virginia Commonwealth University Medical Center (also known as Medical College of Virginia Hospitals) will be eligible for study participation unless they meet study exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study evaluating patients with sepsis is to ascertain differences in cortisol levels between patients with alcohol use disorders and those without alcohol use disorders. | Within 24 hours of hospital admission

SECONDARY OUTCOMES:
A secondary outcome in this study evaluating patients with sepsis is to determine differences in immune function between patients with alcohol use disorders and those without alcohol use disorders. | Within 24 hours of hospital admission
Another secondary aim of this study evaluating patients with sepsis is to determined if higher cortisol levels are associated with increased risk of developing delirium. | Within 72 hours of hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein de Wit, MD, MS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Medical Center (formerly known as Medical College of Virginia), Richmond, Virginia, United States

REFERENCES:
- [Background] O'Brien JM Jr, Lu B, Ali NA, Martin GS, Aberegg SK, Marsh CB, Lemeshow S, Douglas IS. Alcohol dependence is independently associated with sepsis, septic shock, and hospital mortality among adult intensive care unit patients. Crit Care Med. 2007 Feb;35(2):345-50. doi: 10.1097/01.CCM.0000254340.91644.B2. PMID 17205003
- [Background] Moss M, Parsons PE, Steinberg KP, Hudson LD, Guidot DM, Burnham EL, Eaton S, Cotsonis GA. Chronic alcohol abuse is associated with an increased incidence of acute respiratory distress syndrome and severity of multiple organ dysfunction in patients with septic shock. Crit Care Med. 2003 Mar;31(3):869-77. doi: 10.1097/01.CCM.0000055389.64497.11. PMID 12626999
- [Background] de Wit M, Best AM, Gennings C, Burnham EL, Moss M. Alcohol use disorders increase the risk for mechanical ventilation in medical patients. Alcohol Clin Exp Res. 2007 Jul;31(7):1224-30. doi: 10.1111/j.1530-0277.2007.00421.x. Epub 2007 May 20. PMID 17511746
- [Background] de Wit M, Wan SY, Gill S, Jenvey WI, Best AM, Tomlinson J, Weaver MF. Prevalence and impact of alcohol and other drug use disorders on sedation and mechanical ventilation: a retrospective study. BMC Anesthesiol. 2007 Mar 14;7:3. doi: 10.1186/1471-2253-7-3. PMID 17359534
- [Background] Lipiner-Friedman D, Sprung CL, Laterre PF, Weiss Y, Goodman SV, Vogeser M, Briegel J, Keh D, Singer M, Moreno R, Bellissant E, Annane D; Corticus Study Group. Adrenal function in sepsis: the retrospective Corticus cohort study. Crit Care Med. 2007 Apr;35(4):1012-8. doi: 10.1097/01.CCM.0000259465.92018.6E. PMID 17334243
- [Background] Gianoulakis C, Dai X, Brown T. Effect of chronic alcohol consumption on the activity of the hypothalamic-pituitary-adrenal axis and pituitary beta-endorphin as a function of alcohol intake, age, and gender. Alcohol Clin Exp Res. 2003 Mar;27(3):410-23. doi: 10.1097/01.ALC.0000056614.96137.B8. PMID 12658106
- [Background] Kudoh A, Katagai H, Takase H, Takazawa T. Increased cortisol response to surgery in patients with alcohol problems who developed postoperative confusion. Alcohol Clin Exp Res. 2004 Aug;28(8):1187-93. doi: 10.1097/01.alc.0000134229.19493.fc. PMID 15318117
- [Derived] de Wit M, Wiaterek GK, Gray ND, Goulet KE, Best AM, Clore JN, Sweeney LB. Relationship between alcohol use disorders, cortisol concentrations, and cytokine levels in patients with sepsis. Crit Care. 2010;14(6):R230. doi: 10.1186/cc9385. Epub 2010 Dec 22. PMID 21176217